CLINICAL TRIAL: NCT00709917
Title: Observational Study Investigating the Efficacy of Switching From Metformin Monotherapy to a Dual Therapy of Metformin and Repaglinide on Glycaemic Control in Type 2 Diabetes
Brief Title: Observational Study of the Switch of Metformin Alone to Metformin Combined With Repaglinide in Type 2 Diabetes
Acronym: REPAMET
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: AGEE-1857
Record Dates: First submitted 2008-06-30; First posted 2008-07-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: repaglinide

INTERVENTIONS:
Drug: repaglinide — Start dose and freqency to be prescribed by the physician at his discretion following clinical practice
  Other Names: AGEE; Prandin®

SUMMARY:
This study is conducted in Europe.

The aim of this observational study is to investigate the switch from metformin alone to metformin combined with repaglinide in type 2 diabetic patients not achieving adequate glycaemic control on maximal dose of metformin given alone and to analyse different epidemiological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients with inadequate glycaemic control when received metformin alone on maximal dose
* Signed informed consent
* Treatment in accordance with the summary of product characterisation

Exclusion Criteria:

* Any contraindication to metformin or repaglinide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic patients having failed on metformin monotherapy
Sampling Method: Non-Probability Sample
Enrollment: 2171 (Actual)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Safety (number of hypoglycaemic incidents) | After 10-20 weeks
HbA1C | After 10-20 weeks

SECONDARY OUTCOMES:
safety | After 10-20 weeks
posology | After 10-20 weeks
lifestyle | After 10-20 weeks
FBG | After 10-20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Brussels, Belgium
- Luxembourg, Luxembourg

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com